CLINICAL TRIAL: NCT05613374
Title: Virtual Reality-Based Gait Training For Reducing Risk Of Fall in the Elderly.
Brief Title: Gait Training For Reducing Risk Of Fall in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Ehab Mohamed Abd El Kafy, Professor of Physical Therapy, Umm Al-Qura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22UQU4280521DSR01
Record Dates: First submitted 2022-11-05; First posted 2022-11-14 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2022-11

CONDITIONS: Fall
Keywords: The Elderly; Fall Risk; Virtual Reality; Treadmill

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Participants in the control group will receive conventional functional training (conventional physical therapy program) for one hour as the following.
  * Part (1) Postural reactions exercises. (for 30 minutes)
  * Rest for 15 minutes between the first part and the second part.
  * Part (2) Indoor open environment gait training exercises (over-ground gait training exercises.). (for 30 minutes)
  Interventions: Other: Conventional Physical Therapy Program
- Experimental Group (Experimental): Participants in the experimental group will receive a treatment program that is comprised of two parts.
  The first part included training, for (30 minutes), on The C-Mill virtual reality treadmill. The C-Mill is an instrumented treadmill with interactive virtual reality games and applications. The C-Mill applies an augmented virtual reality environment, obstacle avoidance games, and a variety of balance challenges in a safe and controlled environment to increase walking adaptability and performance in everyday life.
  There will be 15 minutes rest between parts one and two of the training program
  The second part (conventional training program) (30 minutes) will include:
  * Postural reactions exercises. ( 20 minutes)
  * Indoor open environment gait training exercises (over-ground gait training exercises.). (10 minutes)
  Interventions: Device: The C-Mill virtual reality treadmill

INTERVENTIONS:
Device: The C-Mill virtual reality treadmill — The C-Mill treadmill is an innovative device used for the training of impaired gait and balance. The C-Mill is an instrumented treadmill with interactive virtual reality games and applications.The instrument is supplied with a safety frame, body weight support, treadmill force plates, treadmill belt, adjustable handrails, cameras, user operating system, interactive visual screen and augmented reality projection.
  Arms: Experimental Group
Other: Conventional Physical Therapy Program — The Conventional Physical Therapy Program include the following:
  * Postural reactions exercises. (using balance board, balance beam, and manual balance perturbations)
  * Indoor open environment gait training exercises (over ground gait training exercises.). (using obstacles,cones , stepper, balance board , and uneven surfaces) (either between or outside the parallel bar)
  Arms: Control Group

SUMMARY:
Falling is considered one of the major problems that may affect the elderly, which may lead to bad consequences. Safe walking needs the older adult to anticipate and respond quickly to external demands and sudden environmental changes.Many studies have shown that treadmill training is effective in improving the elderly person's ability to walk and avoid falls. The C-Mill treadmill is an innovative device that recently used for the training of impaired gait and balance.Therefore, this study will aim to evaluate the efficacy of gait training with a virtual reality treadmill on the risk of fall in the elderly.

DETAILED DESCRIPTION:
Fall injuries produce serious threats to elderly people. Fall hazards are many, they include physical, psychological, social, and economic consequences. Many studies have shown that walking and balance exercises effectively contribute to enhancing walking performance, improving obstacle avoidance, and reducing the incidence of falls in the elderly. Therefore, the practice of complex and challenging situations of the usual daily walking is very important to prevent falls. Many studies have shown that treadmill training is effective in improving the elderly person's ability to walk and avoid falls. The C-Mill treadmill is recently used for the training of impaired gait and balance. C-Mill applies a virtual reality environment, obstacle avoidance games, and a variety of balance challenges in a safe and controlled environment to increase walking adaptability and improve performance in everyday life.Fall injuries produce serious consequences. The management of these injuries is costly and has a negative impact on healthcare entities. Therefore, prevention programs for preventing and reducing falls among the elderly are very important for reducing these serious consequences. Therefore, this study will compare the efficacy of gait training with a virtual reality treadmill and the conventional physical therapy training program on the risk of fall in the elderly.

ELIGIBILITY:
Inclusion Criteria:

60 healthy older adults, both sexes, will participate in this study. Their ages will be between 60 to 70 years. They should have stable medical status based on a confirmed written medical report signed by their physicians. All participants should not receive other training to improve their balance and gait during the duration of the study application except through this study training program.

Exclusion Criteria:

The exclusion criteria will include any participant with:

* a cognitive reduction (< 23 points based on the Mini-Mental State Examination scale;
* muscle paralysis,
* ﬁxed lower limb bony deformities,
* balance deficits,
* visual problems,
* diabetes mellitus,
* polyneuropathy,
* gait disorders,
* using assistive walking devices during walking,
* vertigo, anti-seizures drug use and hypertension,
* vestibular and cerebellar problems; and
* auditory and perceptual diseases/impairments

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Change in the score of fall risk test . (test that assess the change in risk of fall) | [Data will be collected at baseline, and 6 weeks after intervention commencement]
  The Biodex Balance System was used to assess the Change in the Overall Stability Index of the Fall Risk Test. In this study, the dynamic level (11) will be selected for applying the fall risk test. The result for every child will be registered and compared to the normative data stored in the software of the device based on children age range.
Change in the Overall Stability Index {percentage value (%)}, and Time of Control {seconds} for Limit of Stability Test (test that assess the change in balance ability) | [Data will be collected at baseline, and 6 weeks after intervention commencement]
  The Biodex Balance System will be used to assess the change in the Overall Stability Index and the Time of Control of the Limit of Stability Test. This test involves measurement of overall directional control which represented as a percentage value (%). The higher scores will indicate better balance control. The test also include measurement of total time required to complete the test (seconds), improvement in this parameter requires minimizing the time recorded to complete the test.

SECONDARY OUTCOMES:
Change in the Timed Up and Go (TUG) (test that assess the probability for falls among elderly) | [Data will be collected at baseline, and 6 weeks after intervention commencement]
  The Timed Up and Go Test (TUG) will be used to assess the following parameters in older adults: fall risk, walking ability, balance, and mobility. It is a reliable, valid and sensitive test that is a specific measure of the probability for falls among elderly.

CONTACTS AND LOCATIONS:
Overall Officials: Ehab M Abd El Kafy, PhD, Principal Investigator — Department of Physical Therapy- Faculty of Applied Medical Sciences - Umm Al Qura University
Locations (1):
- Ehab Mohamed Abd El Kafy, Mecca, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
- The data available is Case-by-case basis at the discretion of Primary Sponsor
Supporting Information: SAP
Time Frame: Start Date: Beginning one year following main results publication End Date: Ending two years following main results publication
Access Criteria: Data can be obtained by the Principal Investigator. Email Address: emkafy@uqu.edu.sa